CLINICAL TRIAL: NCT03949829
Title: Cardiovascular Disease After Preeclampsia
Brief Title: The CoPenHagen PREeClampsia and cardIOvascUlar diSease Study
Acronym: CPH-PRECIOUS
Status: Active, not recruiting | Type: Observational
Sponsor: Klaus Fuglsang Kofoed (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Klaus Fuglsang Kofoed, Clinical Associated Research Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-18065695
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pre-Eclampsia; Atherosclerosis; Cardiovascular Diseases; Heart Disease in Women
Keywords: Pre- eclampsia; Heart disease in women
MeSH Terms: conditions — Pre-Eclampsia; Atherosclerosis; Cardiovascular Diseases; Toxemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiovascular CT — Cardiac and cardiovascular non-contrast and contrast CT

SUMMARY:
Women with a history of preeclampsia (PE) have increased risk of hypertension and cardiovascular disease (CVD) later in life. Thus, PE is acknowledged as an independent risk factor for CVD, which is the number one cause of death in women in the western part of the world.

Objective:

The purpose of this study is to investigate 1) the prevalence of CVD after PE, 2) which women have the highest risk of developing CVD, 3) when early stages of CVD can be detected in women with previous PE and 4) how CVD progress over time.

Methods:

1000 women with previous PE between the age of 35-55 years will be invited to participate in a follow-up study consisting of anthropometric measurements, blood pressure measurement, urine- and blood samples, cardiac CT-scan and questionnaires. Coronary atherosclerosis will be evaluated using CT imaging.The women will be compared with women with a formerly uncomplicated pregnancy,

Summary:

The study will provide new important information to guide future clinical follow-up, and potentially prevent disease and early death in a large group of women with a history of PE.

DETAILED DESCRIPTION:
Women with a history of preeclampsia (PE) have increased risk of hypertension and cardiovascular disease (CVD) later in life. Thus, PE is acknowledged as an independent risk factor for CVD, which is the number one cause of death in women in the western part of the world. Despite this, solid and uniform guidelines regarding follow-up after a pregnancy complicated by PE are lacking. Little is known about the time-course of the development of CVD and how early stages can be identified in women with previous PE. The link between PE and CVD is well established. However, no large clinical study using cardiac CT-scans exists. Moreover, the study will focus on the time-perspective of the development of CVD in relation to index pregnancy, and this knowledge may prove to be essential to establish solid clinical guidelines addressing timely prevention and treatment.

The purpose of this study is to investigate

1. The prevalence of CVD after PE,
2. Which women have the highest risk of developing CVD
3. When early stages of CVD can be detected in women with previous PE
4. How CVD progress over time.

Thus, we hope to identify a window of opportunity where screening and preventive measures may be relevant and potentially beneficial to these women.

A total of 1000 women with previous PE (aged 35-55 years) will be invited to participate in a clinical follow-up study consisting of anthropometric measurements, blood pressure measurement, urine- and blood samples, cardiac CT-scan (identifying coronary atherosclerotic changes) and questionnaires. These women will be compared to age-matched women, without previous preeclampsia investigated in the Copenhagen General Population Study with an identical CT protocol.

ELIGIBILITY:
Inclusion Criteria

- Women with a history of preeclampsia

Exclusion Criteria

* Severe physical or mental disabilities
* Lack of ability to speak and/or understand Danish language

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: A total of 1000 women with previous preeclampsia will be invited to participate in a post-pregnancy clinical cardiovascular CT follow-up study. These women will be compared to age-matched women, without previous preeclampsia investigated in the Copenhagen General Population Study with an identical CT protocol.
Sampling Method: Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Coronary atherosclerosis | Assessed within 30 days of study inclusion
  Presensence of coronary plaque as defined by Cardiac CT

SECONDARY OUTCOMES:
Presence of left bundle branch block | Assessed within 30 days of study inclusion
  Electrocardiographic abnormality
Presence of atrial fibrillation | Assessed within 30 days of study inclusion
  Electrocardiographic abnormality
Presence of T-wave inversion | Assessed within 30 days of study inclusion
  Electrocardiographic abnormality
Presence of left ventricular hypertrophy | Assessed within 30 days of study inclusion
  Electrocardiographic abnormality
Arterial hypertension | Assessed within 30 days of study inclusion
  Presence of elevated blood pressure
Dyspnoe | Assessed within 30 days of study inclusion
  New York Heart Association class
Chest pain | Assessed within 30 days of study inclusion
  Canadian Cardiovascular Society angina pectoris class

OTHER OUTCOMES:
Major cardiovascular events | Assessed 1 year after Cardiac CT imaging
  Composite endpoint of either death, myocardial infarction, heart failure or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Peter Damm, MD, DmSc, Study Chair — Department of Obstetrics, Rigshospitalet, University of Copenhagen, Denmark
Locations (3):
- Denmark (3):
  - Department of Cardiology and Radiology, Rigshospitalet, The Heart Center, Capital Region of Copenhagen, University of Copenhagen, Copenhagen
  - Department of Obstetrics, Rigshospitalet, Copenhagen
  - The Copenhagen General Population Study, Herlev-Gentofte Hospital, University of Copenhagen, Denmark, Herlev

IPD SHARING:
Plan to Share IPD: Undecided
Logistics and patient data protection issues will be explored prior to decision on IPD

REFERENCES:
- [Derived] Hauge MG, Damm P, Kofoed KF, Moller ELR, Lopez AG, Ersboll AS, Johansen M, Sigvardsen PE, Pham MHC, Goetze JP, Fuchs A, Kuhl JT, Nordestgaard BG, Kober LV, Gustafsson F, Linde JJ. Left Ventricular Hypertrophy in Women With a History of Preeclampsia. Hypertension. 2025 May;82(5):774-783. doi: 10.1161/HYPERTENSIONAHA.124.23497. Epub 2024 Nov 14. PMID 39540300
- [Derived] Hauge MG, Linde JJ, Kofoed KF, Ersboll AS, Johansen M, Sigvardsen PE, Fuchs A, Mikkelsen AP, Gustafsson F, Damm P. Early-onset vs late-onset preeclampsia and risk of coronary atherosclerosis later in life: a clinical follow-up study. Am J Obstet Gynecol MFM. 2024 May;6(5):101371. doi: 10.1016/j.ajogmf.2024.101371. Epub 2024 Apr 6. PMID 38588914
- [Derived] Hauge MG, Damm P, Kofoed KF, Ersboll AS, Johansen M, Sigvardsen PE, Moller MB, Fuchs A, Kuhl JT, Nordestgaard BG, Kober LV, Gustafsson F, Linde JJ. Early Coronary Atherosclerosis in Women With Previous Preeclampsia. J Am Coll Cardiol. 2022 Jun 14;79(23):2310-2321. doi: 10.1016/j.jacc.2022.03.381. PMID 35680182